CLINICAL TRIAL: NCT01732003
Title: The Effect of Omega-3 Fatty Acid Supplementation on Skeletal Muscle Plasma and Mitochondrial Membrane Composition and Cellular Metabolism
Brief Title: The Effect of Omega-3 Fatty Acid Supplementation on Skeletal Muscle Membrane Composition and Cellular Metabolism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Guelph (Other)
Collaborators: McMaster University (Other); Medical University of Bialystok (Other)
Responsible Party: Principal Investigator, Lawrence Spriet, Professor and Chair, University of Guelph
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 11SE032
Record Dates: First submitted 2012-11-17; First posted 2012-11-22 (Estimated); Last update posted 2012-11-28 (Estimated); Status verified 2012-11

CONDITIONS: Skeletal Muscle Energy Metabolism
Keywords: Omega-3; Skeletal Muscle; Eicosapentaenoic acid; Docosahexaenoic acid; Exercise; Membrane Composition; Lipid Metabolism
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omega-3 Complete (Experimental): Oral ingestion of 3000 mg (5 capsules) of Omega-3 Complete (Jamieson Laboratories Ltd., Windsor, Ontario, Canada) per day for 12 weeks
  Interventions: Dietary Supplement: Omega-3 Complete
- Placebo Pill (Placebo Comparator): Oral ingestion of 5 capsules of a placebo oil pill (Jamieson Laboratories Ltd., Windsor, Ontario, Canada) per day for 12 weeks
  Interventions: Dietary Supplement: Placebo Pill

INTERVENTIONS:
Dietary Supplement: Omega-3 Complete
  Arms: Omega-3 Complete
Dietary Supplement: Placebo Pill
  Arms: Placebo Pill

SUMMARY:
The biological membranes that surround a cell and its organelles are vital to the overall function of the cell. Fatty acids are the main structural component of membranes, and the presence of specific fatty acids can alter a membrane's characteristics, which subsequently alters function. Two fatty acids that are of particular interest to researchers are eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA). These omega-3 fatty acids have unique unsaturated structures, and their incorporation into biological membranes appear to elicit potent physiological effects. The body is unable to intrinsically synthesize these important fatty acids, so they must be obtained from the diet or through supplementation.

Compared to research investigating other body tissues, the effect of EPA and DHA on skeletal muscle membranes and cellular function has received little attention. Of the studies done, EPA and DHA supplementation consistently results in increased EPA, DHA, and total omega-3 fatty acid content in the skeletal muscle membranes of rodents. One study has also demonstrated this effect in humans. These studies, however, have been limited to whole muscle measurements, yet cells contain numerous subcellular membranes with diverse functions. Two membranes of key importance to the metabolic function of a skeletal muscle cell are the membrane that surrounds the cell (plasma membrane), and the membrane that surrounds the mitochondria.

The plasma and mitochondrial membranes are responsible for taking up nutrients and converting them into useable energy for the muscle. Recent findings suggest that physiological changes in these processes may occur following EPA and DHA supplementation. At rest and during exercise, there is potential for a shift in substrate selection that favors fat utilization following EPA and DHA supplementation. Several membrane proteins are responsible for transporting fat into the cell and mitochondria. The presence of EPA and DHA within membranes has the potential to affect the membrane integration and function of proteins. The investigators aim to determine whether fat utilization increases following EPA and DHA supplementation, and if there is a concurrent change in the concentrations of fat transport proteins within plasma and mitochondrial membranes. Supplementation with EPA and DHA may also affect oxygen consumption, an important process in energy production that is regulated by mitochondrial membrane proteins. Evidence from human and rodent studies shows a decrease in whole body oxygen consumption following supplementation. The investigators aim to examine these changes directly by measuring mitochondrial respiration following EPA and DHA supplementation.

Therefore, the primary purpose of this study is to examine how plasma and mitochondrial membrane fatty acid composition change individually in response to EPA and DHA supplementation in humans. The secondary purpose of this study is to examine functional metabolic changes that occur in skeletal muscle in response to EPA and DHA supplementation, and to investigate correlational relationships between these changes and any compositional alterations in plasma and mitochondrial membranes. The investigators hypothesize that supplementation with EPA and DHA will alter fuel selection at rest and during exercise, and this will correspond to an increase in the concentration of membrane fatty acid transport proteins, and that these changes will correlate to an increase in the EPA, DHA, and total omega-3 content of plasma and mitochondrial membranes.

ELIGIBILITY:
Inclusion Criteria:

* Recreationally active
* Must currently practice a consistent diet, and exercise regimen, and maintain this throughout the duration of the study

Exclusion Criteria:

* Current or previous supplementation with omega-3s
* Average fish intake greater than two times per week
* Sedentary
* Highly active/trained
* Diagnosed respiratory problem
* Diagnosed heart problem/condition
* Lightheadedness, shortness of breath, chest pain, numbness, fatigue, coughing, or wheezing during at rest of with low to moderate physical activity
* Cardiovascular disease risk factors: Family history of heart attacks, hypertension, hypercholesterolemia, diabetes mellitus, smoking, obesity
* Allergies to lidocaine, fish/fish oil, gelatine, glycerin, or mixed tocopherols
* Currently taking any medications or supplements that may increase the chance of bleeding (e.g. Aspirin, Coumadin, Anti-inflammatories, Plavix, Vitamin C or E, high doses of garlic, ginkgo biloba, willow bark products)
* Tendency toward easy bleeding or bruising

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2011-11; Primary Completion 2013-02 (Estimated); Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
Change in skeletal muscle whole muscle membrane fatty acid composition from baseline | Baseline and 12 weeks
  Percent change in the content of whole muscle membrane fatty acids
Change in skeletal muscle plasma membrane fatty acid composition from baseline | Baseline and 12 weeks
  Percent change in the content of plasma membrane fatty acids
Change in skeletal muscle mitochondrial membrane composition from baseline | Baseline and 12 weeks
  Percent change in the content of mitochondrial membrane fatty acids

SECONDARY OUTCOMES:
Change in whole body resting fat oxidation from baseline | Baseline and 12 weeks
Change in whole body resting carbohydrate oxidation from baseline | Baseline and 12 weeks
Change in whole body sub-maximal exercise fat oxidation from baseline | Baseline and 12 weeks
Change in whole body sub-maximal exercise carbohydrate oxidation from baseline | Baseline and 12 weeks

OTHER OUTCOMES:
Change in resting heart rate from baseline | Baseline and 12 weeks
Change in sub-maximal exercise heart rate from baseline | Baseline and 12 weeks
Change in sub-maximal exercise blood free fatty acid concentration from baseline | Baseline and 12 weeks
Change in sub-maximal exercise blood glucose concentration from baseline | Baseline and 12 weeks
Change in sub-maximal exercise blood lactate concentration from baseline | Baseline and 12 weeks
Change in resting blood C-reactive protein concentration from baseline | Baseline and 12 weeks
Change in resting blood cholesterol concentration from baseline | Baseline and 12 weeks
Change in resting blood high-density lipoprotein concentration from baseline | Baseline and 12 weeks
Change in resting blood low-density lipoprotein concentration from baseline | Baseline and 12 weeks
Change in resting blood cholesterol:high-density lipoprotein ratio from baseline | Baseline and 12 weeks
Change in resting blood triacylglyceride concentration from baseline | Baseline and 12 weeks
Change in resting blood membrane fatty acid content from baseline | Baseline and 12 weeks
Change in skeletal muscle mitochondrial content from baseline | Baseline and 12 weeks
Change in whole muscle fatty acid translocase (FAT/CD36) content from baseline | Baseline and 12 weeks
Change in whole muscle plasma membrane fatty acid binding protein (FABPpm) content from baseline | Baseline and 12 weeks
Change in whole muscle fatty acid transport protein 1 (FATP1) content from baseline | Baseline and 12 weeks
Change in whole muscle fatty acid transport protein 4 (FATP4) content from baseline | Baseline and 12 weeks
Change in whole muscle pyruvate dehydrogenase content from baseline | Baseline and 12 weeks
Change in whole muscle 4-Hydroxynonenal content from baseline | Baseline and 12 weeks
Change in plasma membrane fatty acid translocase (FAT/CD36) content from baseline | Baseline and 12 weeks
Change in plasma membrane fatty acid binding protein (FABPpm) content from baseline | Baseline and 12 weeks
Change in plasma membrane fatty acid transport protein 1 (FATP1) content from baseline | Baseline and 12 weeks
Change in mitochondrial membrane fatty acid translocase (FAT/CD36) content from baseline | Baseline and 12 weeks
Change in mitochondrial respiration from baseline | Baseline and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence L Spriet, PhD, Principal Investigator — University of Guelph
Locations (1):
- University of Guelph, Guelph, Ontario, Canada

REFERENCES:
- [Background] Ayre KJ, Hulbert AJ. Dietary fatty acid profile influences the composition of skeletal muscle phospholipids in rats. J Nutr. 1996 Mar;126(3):653-62. doi: 10.1093/jn/126.3.653. PMID 8598550
- [Background] Peoples GE, McLennan PL. Dietary fish oil reduces skeletal muscle oxygen consumption, provides fatigue resistance and improves contractile recovery in the rat in vivo hindlimb. Br J Nutr. 2010 Dec;104(12):1771-9. doi: 10.1017/S0007114510002928. Epub 2010 Aug 9. PMID 20691135
- [Background] Andersson A, Nalsen C, Tengblad S, Vessby B. Fatty acid composition of skeletal muscle reflects dietary fat composition in humans. Am J Clin Nutr. 2002 Dec;76(6):1222-9. doi: 10.1093/ajcn/76.6.1222. PMID 12450886
- [Background] Couet C, Delarue J, Ritz P, Antoine JM, Lamisse F. Effect of dietary fish oil on body fat mass and basal fat oxidation in healthy adults. Int J Obes Relat Metab Disord. 1997 Aug;21(8):637-43. doi: 10.1038/sj.ijo.0800451. PMID 15481762
- [Background] Delarue J, Labarthe F, Cohen R. Fish-oil supplementation reduces stimulation of plasma glucose fluxes during exercise in untrained males. Br J Nutr. 2003 Oct;90(4):777-86. doi: 10.1079/bjn2003964. PMID 13129446
- [Background] Peoples GE, McLennan PL, Howe PR, Groeller H. Fish oil reduces heart rate and oxygen consumption during exercise. J Cardiovasc Pharmacol. 2008 Dec;52(6):540-7. doi: 10.1097/FJC.0b013e3181911913. PMID 19034030